CLINICAL TRIAL: NCT06087471
Title: Snack Foods and Their Impact on the Gut-Brain Axis: a Randomised Controlled Trial on Mental Health and the Gut Microbiota
Brief Title: Snack Foods and Their Impact on Mental Health and the Gut-brain Axis
Acronym: NutriMood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1423790
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2023-10

CONDITIONS: Depression; Anxiety
Keywords: Mental health; Gut-Brain Axis; Depression; Anxiety; Nutrition; Gut Microbiome
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control snack (Sham Comparator): 42 participants will be randomly assigned to the control snack. Snacks should be consumed twice per day, once as a mid-morning snack and again as a mid-afternoon snack.
  Interventions: Dietary Supplement: Control Snack
- Experimental snack (Experimental): 42 participants (50%) will be randomly assigned to snack on the intervention snack. Snacks should be consumed twice per day, once as a mid-morning snack and again as a mid-afternoon snack.
  Interventions: Dietary Supplement: Intervention snack

INTERVENTIONS:
Dietary Supplement: Intervention snack — The intervention snack will be consumed by 42 participants for 12-weeks. Snacks will be consumed twice a day (mid-morning and mid afternoon snack).
  Arms: Experimental snack
Dietary Supplement: Control Snack — The control snack will be consumed by 42 participants for 12-weeks. Snacks will be consumed twice a day (mid-morning and mid afternoon snack).
  Arms: Control snack

SUMMARY:
The aim of this study is to investigate the effects of snack foods on mental health and the gut-brain axis, in adults with mild to moderate symptoms of depression and anxiety.

DETAILED DESCRIPTION:
There is increasing evidence on the potential modulating role of healthy dietary patterns in managing symptoms of psychological distress including but not limited to depression and anxiety. Despite growing evidence, further research is required to investigate how dietary interventions may impact symptoms of depression and anxiety, as well as their mechanisms of action via the gut-brain axis. Consumption of snacks now contributes to roughly 17% and 21% of daily energy intake for men and women respectively. Therefore, snacks greatly impact nutritional intake and diet quality and can be a target of dietary manipulation for potential health benefits.

This will be the first randomised controlled trial to assess the impact of snack consumption on mental health in adults with mild to moderate symptoms of depression and anxiety. The trial will use a parallel design with a 12-week intervention. Stool and blood samples will be collected at the beginning and end of the intervention for measurement of the gut microbiota and biomarkers related to the gut-brain axis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-45 years old.
* Body mass index (BMI) between 18.50-29.99kg/m2
* Score 10-29 on the patient health questionnaire anxiety and depression scale (PHQ-ADS) for mild to moderate symptoms of depression and anxiety.
* Individuals who regularly consume snacks (Classified as ≥2 per day excluding fruit, vegetable, nut and seed snacks).
* Willing to complete the 12-week intervention by adhering to snacks, complete mental health questionnaires, provide stool and blood samples, record weight and other anthropometric values and record food intake at various timepoints throughout the intervention.
* Willing to adhere to the protocol and provide informed consent.
* Fibre intake of <30g/d
* Willing to discontinue use of pre and probiotics during the trial.

Exclusion Criteria:

* Dislike of intervention products.
* Allergy or intolerance to the intervention products
* Self-report occurrence of substance dependency or severe mental health conditions (e.g., psychosis, schizophrenia, eating disorder). Those with depressive disorders or anxiety disorders will be included in the trial providing they meet all other inclusion criteria.
* Regular consumption of experimental product as snacks and unwilling to complete a washout (no consumption for 4 weeks before baseline or during the study period).
* Changes to medication for depression or anxiety within the last 3 months (e.g., dosage, frequency, type)
* Initiation of any new medications for mental health or any form of talk therapy within the last 3 months.
* Intention to start or alter medication or therapy for mental health during the study.
* Current or previous antibiotic treatment within 4 weeks prior to the start of the study.
* Consumption of probiotics or prebiotic products within the 2 weeks prior to the start of the study
* Women who are pregnant, lactating or planning pregnancy
* Unexplained or unintentional weight loss in the past six months
* Medical history of any of the following: diabetes, major active or historic psychiatric conditions (e.g. schizophrenia), current eating disorder, alcohol abuse, active treatment for cancer in the last year, severe neurological, endocrine, renal, cardiac or pulmonary disease (or any other chronic medical condition), severe oesophagitis, gastritis or duodenitis, active diverticulitis or intestinal/colonic strictures, Coeliac disease, Crohn's disease or Ulcerative colitis, stem cell or organ transplant, gut resection surgery (excluding appendicectomy and cholecystectomy), bleeding disorder, anaphylaxis or any other major or chronic condition known to impact study outcome measures.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Symptoms of depression and anxiety | Week 0 and 12
  Symptoms of depression and anxiety as measured by the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS). This is a 15-item self-report likert scale comprising the PHQ-8 and GAD-7. Scores can range from 0 to 48, cut points of 10,20 and 30 indicate mild, moderate and severe levels of depression/anxiety respectively.

SECONDARY OUTCOMES:
Functional impairment | Weeks 0,6 and 12
  The self-report Work and social adjustment scale (WSAS) will be used to measure functional impairment scores. This is a self-report likert scale with 5 questions. Responses range from Not at all (0) to Very severely (8). 0-9, 10-19 and 20-40 represent low, moderate and severe impairment respectively.
Sleep quality | Weeks 0,6 and 12
  The self-report Pittsburgh sleep quality index (PSQI) will be used to measure sleep quality. This is a 19-item questionnaire with seven subcategories; subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Wellbeing | Weeks 0,6 and 12
  The self-report world health organisation five well-being index (WHO-5) will be used to measure wellbeing. The scale consists of 5 items rated from All of the time (5) to At no time (0).
Quality of life | Weeks 0,6 and 12
  The self-report World Health Organisation Quality of Life Brief (WHOQOL-BREF) scale will be used to measure quality of life. This is a 26-item scale. Responses are rated on a 1-5 likert scale with 1 representing 'not at all' and 5 representing 'completely agree'. Scores are tabulated and multiplied by 4 to represent a score out of 100.
Physical activity | Weeks 0,6 and 12
  The self-report international Physical Activity Questionnaire - Short form (IPAQ) will be used to measure physical activity.
Symptoms of depression | Weeks 0,6 and 12
  The self-report Patient Health Questionnaire-8 (PHQ-8) will be used to measure symptoms of depression. The PHQ-8 is comprised of 8 items rated 0 to 3 with 0 representing 'not at all' and 3 representing 'nearly every day'.
Symptoms of anxiety | Weeks 0,6 and 12
  The self-report Generalised Anxiety disorder-7 scale will be used to measure symptoms of anxiety. The GAD-7 is comprised of 7 questions rated 0 to 3 indicating not at all, to nearly every day respectively.
Psychological Distress | Weeks 0,6 and 12
  The Kessler Psychological Distress Scale (K10) will be used to measure symptoms of psychological distress. The K10 is comprised of 10 questions rated on a 5-point likert scale. Scores range from 10-50.
Faecal gut microbiota (composition, alpha- and beta-diversity) | Week 0 and 12
  Measured by 16S community profiling (Illumina Miseq) of bacterial genomic DNA isolated from stool samples.
Faecal short-chain fatty acids (SCFA) | Week 0 and 12
  Measured by gas liquid chromatography of stool samples
Faecal water | Week 0 and 12
  Determined from stool samples by oven-drying
Gut symptoms | Week 0 and 12
  Measured using the Gastrointestinal Symptom Rating Scale (GSRS) (7-day diary; questionnaire)
Stool frequency | Week 0 and 12
  Measured using self-reported number bowel movements daily recorded in a 7-day diary.
Stool consistency | Week 0 and 12
  Measured using the Bristol stool form scale (7-day dairy; questionnaire)
Serum Vitamin E levels | Week 0 and 12
  Measured in blood sample. Analysis of serum vitamin E levels by Liquid chromatography-mass spectrometry.
Dietary intake | Week 0 and 12
  Measured using a 7-day food and drink diary
Acceptability of snack products | Week 12
  Measured using an Acceptability of dietary intervention questionnaire developed by King's College London for use in dietary intervention studies. The questionnaire assesses acceptability using a number of domains including flavour, texture and portion size.
Snack compliance | Week 12
  Measured via the return of unused snacks at the final visit (consumption of >75% of total snacks will be considered compliant).
Adverse events | Week 0 to 12
  Interview-administered questionnaire
Symptoms of depression and anxiety | Week 0,6 and 12
  Symptoms of depression and anxiety as measured by the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS). This is a 15-item self-report likert scale comprising the PHQ-8 and GAD-7. Scores can range from 0 to 48, cut points of 10,20 and 30 indicate mild, moderate and severe levels of depression/anxiety respectively.
Change in symptoms of depression and anxiety | Week 0, 6 and 12
  Change symptoms of depression and anxiety as measured by the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS). This is a 15-item self-report likert scale comprising the PHQ-8 and GAD-7. Scores can range from 0 to 48, cut points of 10,20 and 30 indicate mild, moderate and severe levels of depression/anxiety respectively.
Proportion of people with no, mild, moderate and severe symptoms of anxiety and depression | Week 0, 6 and 12
  Measured by the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS). This is a 15-item self-report likert scale comprising the PHQ-8 and GAD-7. Scores can range from 0 to 48, cut points of 10,20 and 30 indicate mild, moderate and severe levels of depression and anxiety respectively.
Proportion of people with no, mild, moderate and severe symptoms of depression | Week 0, 6 and 12
  Measured by the PHQ-8 questionnaire. Scores can range from 0 to 24, cut points of 5, 10, 15 and 20 indicate mild, moderate, moderately severe and severe levels of depression, respectively.
Proportion of people with no, mild, moderate and severe symptoms of anxiety | Week 0, 6 and 12
  Measured by the GAD-7. The GAD-7 is comprised of 7 questions rated 0 to 3 indicating not at all, to nearly every day respectively and scores range from 0-21. Cut points are 5, 10 and 15 indicating mild, moderate and severe levels of anxiety, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Metabolic research unit, Franklin-Wilkins Building, 150 stamford street, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No